CLINICAL TRIAL: NCT03547661
Title: Open-Label Placebo Treatment of Women With Premenstrual Syndrome: A Randomized Controlled Trial
Brief Title: Open-Label Placebo Treatment of Women With Premenstrual Syndrome
Acronym: OLPPMS_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Gaab (Other)
Responsible Party: Sponsor-Investigator, Jens Gaab, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 2017-02186; 325130_170117 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2018-05-02; First posted 2018-06-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Open-Label Placebo Effect; randomized controlled trial
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment as Usual (No Intervention): The treatment as usual (TAU) group will control for regression to the mean, spontaneous remission, natural course of disease, and the participants-provider interaction. Participants of the TAU group are allowed to continue their usual medication intake, given they are already on a stable dose (at least 30 days of intake) and the medication is not listed in the exclusion criteria.
- Integrative Open-Label Placebo (Active Comparator): The intervention will encompass an integrative administration of "P-Dragees rosa Lichtenstein", which are pink placebo dragées without any active ingredient. Each dragée contents the following substances: lactose monohydrate; magnesium stearate (Ph. Eur.); microcrystalline cellulose; highly dispersed silicon dioxide; white clay, macrogol glycerolhydroxy stearate (Ph. Eur.); Arabic gum; montanglycol wax; povidone (K 25); talcum; titanium dioxide (E 171); erythrosine; aluminium salt (E 127); calcium carbonate; sucrose; glucose syrup; maize starch; macrogol 6000.
  All participants will be informed that the administered dragées are placebo dragées and participants will be instructed to take two dragées a day for six weeks. (Amendment regarding dosage since 08/18)
  Interventions: Other: P-Dragees rosa Lichtenstein
- Open-Label Placebo (Active Comparator): The intervention will encompass an administration of "P-Dragees rosa Lichtenstein", which are pink placebo dragées without any active ingredient. Each dragée contents the following substances: lactose monohydrate; magnesium stearate (Ph. Eur.); microcrystalline cellulose; highly dispersed silicon dioxide; white clay, macrogol glycerolhydroxy stearate (Ph. Eur.); Arabic gum; montanglycol wax; povidone (K 25); talcum; titanium dioxide (E 171); erythrosine; aluminium salt (E 127); calcium carbonate; sucrose; glucose syrup; maize starch; macrogol 6000.
  All participants will be informed that the administered dragées are placebo dragées and participants will be instructed to take two dragées a day for six weeks. (Amendment regarding dosage since 08/18)
  Interventions: Other: P-Dragees rosa Lichtenstein

INTERVENTIONS:
Other: P-Dragees rosa Lichtenstein — Placebo dragées
  Arms: Integrative Open-Label Placebo; Open-Label Placebo

SUMMARY:
This study aims to investigate the effect of an open-label placebo intervention on premenstrual syndrome (PMS) complaints. Women who suffer from moderate to severe PMS will be randomly allocated to three groups: to a treatment as usual group, an open-label placebo group, and an integrative open-label placebo group. Participants of all groups will conclude a prospective PMS screening for one menstrual cycle. Thereafter, participants of both intervention groups will obtain an openly administered placebo intervention for six weeks. Participants of the treatment as usual group will have the chance to obtain the same open-label placebo intervention after study conduct. Diverse measures will be assessed by means of a PMS symptom diary and questionnaires. Furthermore, we assess participants experiences of study participation qualitatively by means of semi-structured interviews.

DETAILED DESCRIPTION:
Recent evidence suggests that in certain clinical conditions - such as chronic low-back pain, migraine, irritable bowel syndrome, attention deficit hyperactivity disorder, and rhinitis - placebos improve clinical outcomes even without deception. Premenstrual syndrome (PMS) is defined as clinically significant symptoms, comprising at least one emotional or physical symptom in the premenstrual phase of the menstrual cycle and which cause substantial distress or functional impairment. To date, there exists no study examining open-label placebo responses on PMS. However, PMS seems to be considerably susceptible to placebo effects: The Royal College of Obstetricians and Gynaecologists alerts to substantial placebo responses in randomized-controlled PMS trials and studies showed considerable placebo effects on PMS without any specific effect for the medication under examination. Furthermore, a myriad of distinctive therapies is described for PMS (including pharmacological and phytopharmaceutical drugs as well as complementary non-pharmacological interventions), yet partially mixed evidence is reported. Besides being considered as placebogenic, PMS symptoms are timely well-defined and delimited which further makes this condition attractive for an investigation of open-label placebo responses, as a possible amelioration can be measured in a delimited time frame. To sum up, a randomized controlled trial of an open-label placebo treatment of women with PMS allows to investigate ways to harness placebo effects ethically in clinical practice for syndromes with somatic and psychologically described characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe PMS
* Between 18 and 45 years of age
* A regular menstrual cycle, i.e., max. +/- 3 days of difference of cycle range
* Menstrual cycle range not longer than 31 or shorter than 24 days
* Participants have a general practioner or gynaecologist to consult
* At least one premenstrual symptom causes the desire for a PMS treatment

Exclusion Criteria:

* Brest feeding at the moment or during the last three months
* Pregnancy
* Failing menstruation onset in the course of two consecutive menstrual cycles
* An essential mental or somatic disease
* Drug or massive alcohol intake or of other psychoactive substances
* Uptake of a new medication within the last 30 days
* Menopause, premenopausal strain or amenorrhoea
* Allergy of one of the ingredients of the placebo dragées (P-Dragees rosa Lichtenstein)
* Women who are surgically sterilised, hysterectomised, or ovariectomised
* BMI above 30
* Actual or recent participation in psychotherapy due to premenstrual symptoms
* Parallel participation in another study with investigational drugs or participation in another PMS study within the last three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
PMS symptom intensity assessed by a PMS symptom diary sub sum score | Continuous measurement, starting from day 1 of the menstrual cycle (length of each cycle is on average 28 days) until the individual last day of the third menstrual cycle of each participant (assessment across three menstrual cycles in total)
  Symptom intensity will be assessed by an intensity sub scale of the PMS symptom diary. Intensity will be rated by means of a six-level Likert scale, whereat 1 is the lowest rating of symptom intensity and 6 the highest.
PMS symptom interference assessed by a PMS symptom diary sub sum score | Continuous measurement, starting from day 1 of the menstrual cycle (length of each cycle is on average 28 days) until the individual last day of the third menstrual cycle of each participant (assessment across three menstrual cycles in total)
  Symptom interference will be assessed by an interference sub scale of the PMS symptom diary. Interference will be rated by means of a six-level Likert scale, whereat 1 is the lowest rating of interference and 6 the highest.

SECONDARY OUTCOMES:
Experience of study participation in intervention groups | One time assessment, up to 2 years after baseline. The interview takes between 30 and 60 minutes
  By means of semi-structured interviews, participants experience of participation in interventions groups of 10 women of the open-label placebo without treatment rationale group and of 10 women of the open-label placebo with treatment rationale group, who are randomly chosen out of the 50 participants of each of the intervention study groups will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof. Dr., Principal Investigator — University of Basel, Faculty of Psychology, Division for Clinical Psychology and Psychotherapy
Locations (1):
- University of Basel, Faculty of Psychology, Division of Clinical Psychology and Psychotherapy, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho C, Caetano JM, Cunha L, Rebouta P, Kaptchuk TJ, Kirsch I. Open-label placebo treatment in chronic low back pain: a randomized controlled trial. Pain. 2016 Dec;157(12):2766-2772. doi: 10.1097/j.pain.0000000000000700. PMID 27755279
- [Background] Kam-Hansen S, Jakubowski M, Kelley JM, Kirsch I, Hoaglin DC, Kaptchuk TJ, Burstein R. Altered placebo and drug labeling changes the outcome of episodic migraine attacks. Sci Transl Med. 2014 Jan 8;6(218):218ra5. doi: 10.1126/scitranslmed.3006175. PMID 24401940
- [Background] Kaptchuk TJ, Friedlander E, Kelley JM, Sanchez MN, Kokkotou E, Singer JP, Kowalczykowski M, Miller FG, Kirsch I, Lembo AJ. Placebos without deception: a randomized controlled trial in irritable bowel syndrome. PLoS One. 2010 Dec 22;5(12):e15591. doi: 10.1371/journal.pone.0015591. PMID 21203519
- [Background] Maharaj S, Trevino K. A Comprehensive Review of Treatment Options for Premenstrual Syndrome and Premenstrual Dysphoric Disorder. J Psychiatr Pract. 2015 Sep;21(5):334-50. doi: 10.1097/PRA.0000000000000099. PMID 26352222
- [Background] O'Brien, P. S., Rapkin, A., & Schmidt, P. J. (2007). The premenstrual syndromes: PMS and PMDD: CRC Press.
- [Background] Sampson GA. Premenstrual syndrome: a double-blind controlled trial of progesterone and placebo. Br J Psychiatry. 1979 Sep;135:209-15. doi: 10.1192/bjp.135.3.209. PMID 385093
- [Background] Sandler AD, Bodfish JW. Open-label use of placebos in the treatment of ADHD: a pilot study. Child Care Health Dev. 2008 Jan;34(1):104-10. doi: 10.1111/j.1365-2214.2007.00797.x. PMID 18171451
- [Background] Schaefer M, Harke R, Denke C. Open-Label Placebos Improve Symptoms in Allergic Rhinitis: A Randomized Controlled Trial. Psychother Psychosom. 2016;85(6):373-374. doi: 10.1159/000447242. Epub 2016 Oct 15. No abstract available. PMID 27744433
- [Background] Van Ree JM, Schagen Van Leeuwen JH, Koppeschaar HP, Te Velde ER. Unexpected placebo response in premenstrual dysphoric disorder: implication of endogenous opioids. Psychopharmacology (Berl). 2005 Oct;182(2):318-9. doi: 10.1007/s00213-005-0090-8. Epub 2005 Oct 19. No abstract available. PMID 16001107
- [Background] Yonkers KA, O'Brien PM, Eriksson E. Premenstrual syndrome. Lancet. 2008 Apr 5;371(9619):1200-10. doi: 10.1016/S0140-6736(08)60527-9. PMID 18395582
- [Background] Frey Nascimento A, Gaab J, Degen B, Rytz M, Holder A, Sezer D, Buergler S, Meyer AH, Kirsch I, Kossowsky J, Locher C. Efficacy of open-label placebos for premenstrual syndrome: a randomised controlled trial. BMJ Evid Based Med. 2025 Mar 25;30(5):295-304. doi: 10.1136/bmjebm-2024-112875. Online ahead of print. PMID 40132912
- [Derived] Frey Nascimento A, Gaab J, Kirsch I, Kossowsky J, Meyer A, Locher C. Open-label placebo treatment of women with premenstrual syndrome: study protocol of a randomised controlled trial. BMJ Open. 2020 Feb 17;10(2):e032868. doi: 10.1136/bmjopen-2019-032868. PMID 32071176